CLINICAL TRIAL: NCT03862339
Title: UltraSOUND-based Characterization of Ventricular Tachycardia SCAR and Arrhythmogenic Substrate; The SOUNDSCAR Study
Brief Title: The SoundScar Study The SOUNDSCAR Study
Acronym: SoundScar
Status: Completed | Type: Observational
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1171
Record Dates: First submitted 2019-02-25; First posted 2019-03-05 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Ventricular Tachycardia; Ischemic Cardiomyopathy
Keywords: Catheter Ablation
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, Non-randomized, Single-arm Study to assess the accuracy of intracardiac echocardiography (ICE) for characterization of arrhythmogenic substrate in patients with ischaemic cardiomyopathy undergoing ventricular tachycardia (VT) ablation

DETAILED DESCRIPTION:
ICE imaging during VT ablation is currently largely used for definition of cardiac anatomy. The role of the technique to specifically define scar and arrhythmogenic substrate has not been systematically evaluated. The aim is to assess the efficacy of the technique to accurately define the arrhythmogenic substrate.

ELIGIBILITY:
Inclusion Criteria:

* Prior heart attack (myocardial infarction) with evidence from prior non-invasive imaging demonstrating regions of the heart with reduced heart muscle function (myocardial hypokinesia/akinesia/thinning) in the absence of a non-heart attack-related (non-ischaemic) cause
* Age over 18 years
* One of the following abnormal heart rhythm (VT) events within last 6 months:
* ≥3 episodes of VT treated with therapeutic rapid pacing from an implantable cardiac defibrillator (antitachycardia pacing [ATP])
* ≥1 appropriate shocks from an implantable cardiac defibrillator
* ≥3 episodes of abnormal heart rhythm (VT) within 24 hours
* Sustained VT below the detection rate of the implantable cardiac defibrillator (documented by ECG/cardiac monitor)
* Sustained abnormal heart rhythm (VT) in the absence of ICD which is documented by ECG/cardiac monitor
* Patients in whom ICE imaging is planned for the clinical VT ablation procedure (clinical indication)

Exclusion Criteria:

* Patient unable or unwilling to provide informed consent.
* Acute heart attack (acute coronary syndrome with acute thrombus diagnosed by coronary angiography, or dynamic ST segment changes demonstrated on ECG) or another reversible cause of abnormal heart rhythm (VT) - e.g. electrolyte abnormalities or drug-induced abnormal heart rhythms
* Ineligible for ablation (known to have protruding clot in the chamber of interest (left ventricular thrombus), or have implanted mechanical aortic and mitral valves)
* Had recent coronary bypass surgery (< 3 months) or percutaneous coronary intervention (<3 months)
* Pregnant patients (pregnancy test will be performed in patients who are of childbearing age who are not on an effective contraceptive prior to all VT ablation procedures)
* Had recent coronary bypass surgery (< 3 months) or percutaneous coronary intervention (<3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischaemic cardiomyopathy undergoing ventricular tachycardia (VT) ablation
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Areas of abnormal contraction (hypokinesia/akinesia) as determined by ICE imaging | 1 week
  Area with abnormal contraction as correlated the findings on voltage mapping (low voltage) of the left ventricle in patients with a prior myocardial infarction undergoing VT ablation.

SECONDARY OUTCOMES:
Areas of abnormal contraction as determined by ICE imaging | 1 week
  Area of abnormal contraction correlating with the findings on voltage mapping (local abnormal ventricular activities) of the left ventricle in patients with a prior myocardial infarction undergoing VT ablation

CONTACTS AND LOCATIONS:
Overall Officials: Saagar Mahida, MD, Principal Investigator — Liverpool Heart and Chest Hospital; Sharad Agarwal, MD, Principal Investigator — Papworth Hospital NHS Trust
Locations (2):
- Westmead Hospital, Sydney, New South Wales, Australia
- Liverpool Heart and Chest Hospital NHS Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No